CLINICAL TRIAL: NCT02699060
Title: Experimental Study to Determine the Effects of Human Refluxate (Biliary, Gastric, Duodenogastric) on Macrophage Phenotype and Its Correlation With Different Forms of GERD: Motility Talent Group Study
Brief Title: Experimental Study to Determine the Effects of Human Refluxate on Macrophage Phenotype and Its Correlation With GERD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ivashkin Vladimir Trofimovich (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor-Investigator, Ivashkin Vladimir Trofimovich, MD, PhD, professor, head of department of propedeutics of internal diseases, director of clinic of propedeutics of internal diseases, I.M. Sechenov First Moscow State Medical University
Organization: I.M. Sechenov First Moscow State Medical University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EPIDKO19
Record Dates: First submitted 2016-02-12; First posted 2016-03-04 (Estimated); Results first posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: GERD; Barrett's esophagus; macrophage; FSSG questionnaire
MeSH Terms: conditions — Gastroesophageal Reflux; Barrett Esophagus | interventions — Endoscopy, Digestive System; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- NERD patients (Experimental): Patients have typical reflux syndrome without esophageal injury.
  Interventions: Procedure: Upper gastrointestinal endoscopy with biopsy and collection of refluxate; Procedure: Esophageal high-resolution manometry and 24-h esophageal pH-impedance monitoring
- EE patients (Experimental): Patients have erosion(s) or ulcer(s) in esophagus.
  Interventions: Procedure: Upper gastrointestinal endoscopy with biopsy and collection of refluxate; Procedure: Esophageal high-resolution manometry and 24-h esophageal pH-impedance monitoring
- BE patients (Experimental): Patients have esophageal specialized intestinal metaplasia.
  Interventions: Procedure: Upper gastrointestinal endoscopy with biopsy and collection of refluxate; Procedure: Esophageal high-resolution manometry and 24-h esophageal pH-impedance monitoring

INTERVENTIONS:
Procedure: Upper gastrointestinal endoscopy with biopsy and collection of refluxate — we analyzed esophageal mucosa, expression of inflammatory changes, location, size, number of mucosal defects, as well as the appearance of the gastric and duodenal mucosa.
  Other Names: EGD (esophagogastroduodenoscopy) with esophagus biopsy
Procedure: Esophageal high-resolution manometry and 24-h esophageal pH-impedance monitoring — we analyzed following HRM parameters: the distal contractile integral (DCI), the lower esophageal sphincter resting pressure (LES RP) and standard measuring parameters were be collected: percentage of total time when pH was <4, longest reflux event, number of reflux events longer than 5 minutes, and number of reflux episodes in 24 hours.
  Other Names: HRM and 24-h esophageal pH monitoring

SUMMARY:
This study is proposed to evaluate the role of motoric dysfunctions and type of refluxate in GERD patients, analyzed the blood monocyte/macrophage phenotypes of gastroesophageal reflux diseases (GERD) patients.

DETAILED DESCRIPTION:
Patients with non-erosive gastroesophageal reflux disease (NERD), erosive esophagitis (EE) and Barrett esophagus (BE) were enrolled. We investigated blood monocyte/macrophage phenotype in patients with different forms of GERD. We analysed of macrophages phenotype by CD25, CD80, CD163, CD206 expression for M2 macrophages. All patients underwent upper gastrointestinal endoscopy with esophagus biopsy. GERD patients underwent esophageal high-resolution manometry (HRM) with a 22-channel water-perfused catheter and Solar GI system (Medical Measurements Systems, Enschede, the Netherlands) and 24-hour impedance and pH monitoring using the Ohmega Ambulatory Impedance pH Recorder (Medical Measurements Systems).

ELIGIBILITY:
Inclusion Criteria:

Clinical (patients) part

1. Signed informed consent
2. Gender: Male or Female
3. Age: 18-65 years of age

3. Clinically and/or endoscopically confirmed diagnosis of GERD

Exclusion Criteria:

Clinical: (patient)

1. Current treatment with proton pump inhibitors and/or histamine-2 receptor antagonists. These treatments should have been stopped at least 1 week prior to study inclusion.
2. Female patients who are pregnant, planning to become pregnant or lactating
3. Any acute diseases or conditions, exacerbations of concomitant chronic diseases (including but not limited to inflammatory bowel disease (IBD), ulcer disease etc.) at study start/inclusion and/or which are not resolved 14 days prior to study-enrolment.
4. Participation in a clinical trial in the past 3 months
5. Any condition which, in the opinion of investigator, makes the patient unsuitable for participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-02; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Ivashkin, MD,PhD,Prof., Principal Investigator — I.M. Sechenov First Moscow State Medical University
Locations (2):
- Russia (2):
  - I.M.Sechenov First Moscow State Medical University, Moscow
  - Moscow State University of Medicine and Dentistry named after A.I. Evdokimov, Moscow

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhong YQ, Lin Y, Xu Z. Expression of IFN-gamma and IL-4 in the esophageal mucosa of patients with reflux esophagitis and Barrett's esophagus and their relationship with endoscopic and histologic grading. Dig Dis Sci. 2011 Oct;56(10):2865-70. doi: 10.1007/s10620-011-1696-9. Epub 2011 Apr 9. PMID 21479676
- [Background] Kohata Y, Fujiwara Y, Machida H, Okazaki H, Yamagami H, Tanigawa T, Watanabe K, Watanabe T, Tominaga K, Wei M, Wanibuchi H, Arakawa T. Role of Th-2 cytokines in the development of Barrett's esophagus in rats. J Gastroenterol. 2011 Jul;46(7):883-93. doi: 10.1007/s00535-011-0405-y. Epub 2011 May 18. PMID 21590343
- [Background] Gough MD, Ackroyd R, Majeed AW, Bird NC. Prediction of malignant potential in reflux disease: are cytokine polymorphisms important? Am J Gastroenterol. 2005 May;100(5):1012-8. doi: 10.1111/j.1572-0241.2005.40904.x. PMID 15842572
- [Background] Fitzgerald RC, Onwuegbusi BA, Bajaj-Elliott M, Saeed IT, Burnham WR, Farthing MJ. Diversity in the oesophageal phenotypic response to gastro-oesophageal reflux: immunological determinants. Gut. 2002 Apr;50(4):451-9. doi: 10.1136/gut.50.4.451. PMID 11889061
- See also: I.M.Sechenov First Moscow State Medical University website — http://www.mma.ru/en/

RESULTS

PARTICIPANT FLOW:
Groups:
- GERD: NERD patients, EE patients and BE patients
Period: Overall Study
Arm/Group | GERD
Started | 68
Completed | 68
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: participants
Groups:
- Non Erosive Reflux Disease; Erosive Esophagitis; Barrett's Esophagus: Participants not received drugs
- Total: Total of all reporting groups
Arm/Group | Non Erosive Reflux Disease | Erosive Esophagitis | Barrett's Esophagus | Total
Number analyzed (Participants) | 28 | 22 | 18 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] — years
  years | 45.74 (2.23) | 45.0 (3.24) | 47.22 (2.95) | 46.8 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 7 | 5 | 26
  Male | 14 | 15 | 13 | 42
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 28 | 22 | 18 | 68
Expression levels macrophage CD markers from GERD patients [Mean (Standard Deviation); unit: mg/l]
  CD25 | 34.6 (15.9) | 34.2 (14.0) | 40.0 (14.4) | 36.9 (15.2)
  CD80 | 23.0 (13.3) | 23.5 (10.0) | 24.4 (11.5) | 23.4 (11.8)
  CD163 | 16.6 (15.9) | 18.0 (10.0) | 14.3 (8.1) | 16.3 (9.1)
  CD206 | 10.4 (7.2) | 11.9 (8.0) | 9.6 (7.7) | 10.6 (7.5)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Reflux in GERD Patients
Description: We analyzed the number of acid and weakly acid reflux episodes in GERD patients
Time Frame: Day 4
Measure: Median (Inter-Quartile Range); unit: episodes
Groups:
- NERD Patients: Patients with heartburn were found to exhibit inflammatory esophageal mucosa during endoscopy
- EE Patients: Patients with erosions or ulcers in esophagus by endoscopy
- BE Patients: Patients with intestinal metaplasia in esophagus
Arm/Group | NERD Patients | EE Patients | BE Patients
Number analyzed (Participants) | 28 | 22 | 18
episodes
  The acid reflux episodes | 33.6 [0 to 79.0] | 42.8 [2.0 to 111.0] | 81.0 [12.0 to 211.0]
  The weakly acid reflux episodes | 53.1 [28.8 to 99.0] | 34.4 [12.0 to 100.0] | 31.8 [4.0 to 100.0]
Statistical Analysis 1: Comparison: NERD Patients vs EE Patients vs BE Patients; Test type: Superiority; p = 0.002, Mixed Models Analysis; Median Difference (Net) = -1.76, Standard Deviation 0.80

ADVERSE EVENTS:
Time Frame: 32 weeks
Description: We haven't adverse events because we not used drugs in our study.
Groups:
- NERD Patients: Patients have the typical reflux syndrome without esophageal injury.
- BE Patients: Patients have specialized esophageal intestinal metaplasia.
Arm/Group | NERD Patients | EE Patients | BE Patients
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/22 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/22 | 0/18
Other Adverse Events (participants affected / at risk) | 0/28 | 0/22 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-12): https://cdn.clinicaltrials.gov/large-docs/60/NCT02699060/Prot_SAP_000.pdf